CLINICAL TRIAL: NCT01685554
Title: Normothermiс Cardiopulmonary Bypass Increases Cerebral Oxygenation During Combined Valve Surgery: Single Center, Randomized Trial
Brief Title: Normothermiс Cardiopulmonary Bypass Increases Cerebral Oxygenation During Valve Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Norm-Arh-2012
Record Dates: First submitted 2012-09-04; First posted 2012-09-14 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Heart Valve Diseases
Keywords: perfusion; cardiopulmonary bypass; hypothermia; cerebral oxygenation
MeSH Terms: conditions — Heart Valve Diseases; Hypothermia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- normothermic CPB (Active Comparator): cardiopulmonary bypass with maintenance of normal body temperature
  Interventions: Device: normothermic CPB
- hypothermic CPB (Active Comparator): cardiopulmonary bypass using mild hypothermia
  Interventions: Device: hypothermic CPB

INTERVENTIONS:
Device: hypothermic CPB — maintenance of mild hypothermia during cardiopulmonary bypass
  Arms: hypothermic CPB
Device: normothermic CPB — maintenance of normal body temperature during cardiopulmonary bypass
  Arms: normothermic CPB

SUMMARY:
The aim of our study was to evaluate the effect of different temperature regimens of cardiopulmonary bypass on systemic oxygen transport and cerebral oxygenation during surgical correction of acquired heart diseases.

DETAILED DESCRIPTION:
Our aim was to evaluate the effect of hypothermic and normothermic regimens of cardiopulmonary bypass on systemic oxygen transport and cerebral oxygenation during valve surgery

ELIGIBILITY:
Inclusion Criteria:

* requirement of surgical correction of two or more valves

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Cerebral oxygen saturation | perioperatively
  measurement of cerebral oxygen saturation during cardiopulmonary bypass and 24 hrs postoperatively

SECONDARY OUTCOMES:
time until "fit for ICU discharge" fulfillment | 5 days postoperatively
  measurement of time to fulfillment of the "fit for discharge" criteria

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Y Kirov, MD, PhD, Study Director — Northern State Medical Univercity
Locations (1):
- Dep. of Anesthesiology, Northern SMU, Arkhangelsk, Russia

REFERENCES:
- [Derived] Lenkin AI, Zaharov VI, Lenkin PI, Smetkin AA, Bjertnaes LJ, Kirov MY. Normothermic cardiopulmonary bypass increases cerebral tissue oxygenation during combined valve surgery: a single-centre, randomized trial. Interact Cardiovasc Thorac Surg. 2013 May;16(5):595-601. doi: 10.1093/icvts/ivt016. Epub 2013 Feb 13. PMID 23407696